CLINICAL TRIAL: NCT04085692
Title: Dispatcher-Assisted Cardiopulmonary Resuscitation: A Randomized Controlled Trial of Low-Dose, High-Frequency Simulation-Based Training and the Impact on Real Out-of-Hospital Cardiac Arrest Calls
Brief Title: Dispatcher-Assisted CPR: Low-Dose, High-Frequency Simulation-Based Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emergency Medical Services, Capital Region, Denmark (Other Government)
Collaborators: TrygFonden, Denmark (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: DTP
Record Dates: First submitted 2019-09-02; First posted 2019-09-11 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Out-Of-Hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Intervention Model Description: After enrolment and consent from the EMDs, the EMDs will be randomly assigned to receive either LDHF simulation-based dispatcher training (intervention arm) or no LDHF simulation-based dispatcher training (comparison arm).
  The EMDs will be randomly assigned to intervention or comparison group in a 1:1 ratio.
  Randomisation will be stratified by the EMDs' medical backgrounds (paramedic, approximately 30% of the EMDs, or registered nurse, approximately 70% of the EMDs), to balance the number of EMDs with different medical backgrounds randomly assigned to each arm.
Who Masked: Outcomes Assessor
Masking Description: The research group and the participants will not be blinded to the allocation, except for the study statistician (A.K.E.), who will conduct all analyses blinded to the intervention group. Thus, the study statistician will not have access to the randomisation scheme or the random seed and will receive a dataset with the actual groups replaced with the numbers 0 and 1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group begins LDHF dispatcher training with one introduction week followed by twelve weeks of LDHF training.
  During the study period, all regular quality improvement (QI) activities, such as self-audits, case reviews, mentor groups, and status meetings will continue for all EMDs.
  Interventions: Behavioral: Low-Dose, High-Frequency Simulation-Based Training
- Comparison (No Intervention): During the study period, all regular quality improvement (QI) activities, such as self-audits, case reviews, mentor groups, and status meetings will continue for all EMDs.

INTERVENTIONS:
Behavioral: Low-Dose, High-Frequency Simulation-Based Training — Twelve weeks of LDHF training
  The simulation-based training sessions take place at the EMDC, at extra workstations set-up as ordinary EMD workstations in an out-of-the-way area. Before each session, the EMD is informed about the simulation call and receives instructions concerning technical differences from a regular call. The instructor acts as a "standardised caller", guided by a computer program. This program, the Danish version of Resuscitation Quality Improvement for Telecommunicators (Laerdal Medical AS, Stavanger, Norway), is a training program for DA-CPR based on the simulation platform Laerdal Learning Application. This modified version of the RQI-T program has, one test scenario, one data collection scenario and six different cardiac arrests scenarios as well as a feedback checklist based on the Danish dispatcher protocol Danish Index for Emergency Care.
  Each simulation session takes approximately 20 minutes, including introduction and feedback
  Arms: Intervention

SUMMARY:
Clear, concise, yes, and no answers can be challenging to achieve in the assessment of consciousness and breathing in out-of-hospital cardiac arrest (OHCA) calls. Often callers will provide an unclear response, and this can lead to hesitation on the part of the Emergency Medical Dispatcher (EMD). Further, the relatively small proportion OHCA calls represent might demand the need for simulation training in the dispatcher-assisted cardiopulmonary resuscitation (DA-CPR) guiding itself. Therefore, the investigators investigate whether low-dose, high-frequency (LDHF) simulation-based training of EMDs can increase the quality of DA-CPR in a simulation setting. Additionally, the investigators measure whether the effect of the training will be transferred to real OHCA calls.

The study is a randomised controlled trial comparing LDHF simulation-based training to standard quality improvement of the EMD in a single centre. The study protocol is structured according to the SPIRIT 2013 statement, and the study will be reported in compliance with the CONSORT 2010 Statement. The investigators chose EMDs receiving standard quality improvement as the comparator group, to reflect a representative cohort of the EMDs not exposed to the LDHF simulation-based training program.

The aims of this study are:

1. To measure the effect of LDHF simulation-based training on the quality of DA-CPR in a simulation setting.
2. To measure the effect of LDHF simulation-based training on the quality of DA-CPR in real OHCA calls.

The investigators hypothesise that LDHF simulation-based training will increase the quality of DA-CPR in the intervention group in a simulation setting and that this improvement is transferred to real OHCA calls - although the effect in real OHCA calls might be smaller due to the complexity of some calls. The investigators hypothesise that this improvement can be detected as a decrease in time to first bystander compression (TTFC), an increase in clarification of consciousness and breathing without asking additional questions, a decrease in time to recognition of cardiac arrest, and an increase in calls where the EMD provide DA-CPR instructions on patients in cardiac arrest.

ELIGIBILITY:
Inclusion criteria:

- EMD employed at the Copenhagen EMS at the time of enrolment.

Exclusion criteria:

* Mean working time as call taker at Copenhagen EMS < 8 hours/week.
* Planned employment cessation at the Copenhagen EMS during the data collection period.
* Planned leave from work longer than four weeks during the data collection period.
* Starting employment at the Copenhagen EMS during the study period.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2019-12-25 (Actual); Study Completion 2019-12-25 (Actual)

PRIMARY OUTCOMES:
Time from a call is taken by EMD to first bystander compression | During cardiac arrest calls, up to 1 hour
  (seconds)

SECONDARY OUTCOMES:
EMD clarifies status of consciousness and breathing before asking any additional questions | During cardiac arrest calls, up to 1 hour
  (yes/no)
Time from a call is taken by EMD to the recognition of cardiac arrest | During cardiac arrest calls, up to 1 hour
  (seconds)
EMD starts DA-CPR instructions | During cardiac arrest calls, up to 1 hour
  (yes/no)
Time from a call is taken by EMD to EMD starts DA-CPR instructions | During cardiac arrest calls, up to 1 hour
  (seconds)
EMD is assertive when starting CPR instructions | During cardiac arrest calls, up to 1 hour
  (yes/no)
EMD starts DA-CPR instructions on patient without cardiac arrest | During cardiac arrest calls, up to 1 hour
  (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Freddy Lippert, MD, Principal Investigator — Emergency Medical Services, Capital Region, Denmark; Oscar Rosenkrantz, Study Director — Emergency Medical Services, Capital Region, Denmark
Locations (1):
- Copenhagen Emergency Medical Services, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Immediately following publication. Until 31st of December 2021
Access Criteria: Researchers who provide a sound proposal and gets approval from the Danish authorities.

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: Full protocol (2019-09-02): https://cdn.clinicaltrials.gov/large-docs/92/NCT04085692/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-05): https://cdn.clinicaltrials.gov/large-docs/92/NCT04085692/ICF_001.pdf
  • Study Protocol: Supplementary assessment points for table 1 (2019-12-27): https://cdn.clinicaltrials.gov/large-docs/92/NCT04085692/Prot_002.pdf